CLINICAL TRIAL: NCT01351597
Title: An Open-label, Multi-center Phase II Trial to Evaluate the Efficacy and Safety of Combination Chemotherapy With DoceTaxel(Detaxel) and Oxaliplatin(Oxalitin)in Recurrent or Metastatic Breast Cancer
Brief Title: A Clinical Trial of Docetaxel and Oxaliplatin in Patients With Recurrent or Metastatic Breast Cancer
Acronym: STORM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean Breast Cancer Study Group (Other)
Responsible Party: Sehwan Han, Department of Surgery, Breast Cancer Center, Inje University Paik Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KBCSG008
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Recurrent Breast Cancer; Metastatic Breast Cancer
Keywords: recurrent breast cancer; metastatic breast cancer; docetaxel; oxaliplatin
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- docetaxel/ oxaliplatin (Experimental): All the patients are recurrent or metastatic breast cancer. Patients with a measurable lesion.
  Interventions: Drug: docetaxel/ oxaliplatin

INTERVENTIONS:
Drug: docetaxel/ oxaliplatin — 1. docetaxel - 75 mg/m2 with D5W250ml IV (in the vein)over 1 hr, every 3 weeks
  2. oxaliplatine - 70 mg/m2 with D5W250ml IV (in the vein)over 2 hrs, every 3 weeks
  Other Names: Detaxel®; oxalitin®

SUMMARY:
The purpose of this study is to evaluate the overall response rate, toxicity, progression free survival and quality of life of chemotherapy with docetaxel and oxaliplatin in recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
Recent therapeutic developments, such as the introduction of new cytotoxic agents (taxanes, platinum, liposomal anthracyclines, etc) have resulted in constant improvements in treatment efficacy and consequently in recurrent or metastatic outcome. This single arm, multicenter phase II study was designed to evaluate the response rate, toxicity, progression free survival of docetaxel and oxaliplatin in patients with recurrence or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged : 20~70 years
2. WHO (ECOG) performance status 0-2
3. Patients with measurable lesion assessed by imaging using the RECIST (Response Evaluation Criteria In Solid Tumor) guideline
4. patients had previously not received chemotherapy of recurrent or metastatic lesion.
5. Have given written informed consent and are available for prolonged follow-up

Exclusion Criteria:

1. Patients with previous chemotherapy for recurrent breast cancer
2. Breast cancer recurrence within 12 months after taxane treatment
3. Her-2/neu expression breast cancer
4. Patients with malignancies (other than breast cancer) within the last 5 years, except for adequately treated in situ carcinoma of the cervix or basal cell, squamous cell carcinoma of the skin.
5. Brain metastasis
6. uncontrolled infection, medically uncontrollable heart disease
7. other serious medical illness or prior malignancies
8. Pregnant or lactating women were excluded.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 2 years

SECONDARY OUTCOMES:
progression free survival | 2 years
toxicity | 2 years
quality of life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sehwan Han, MD.PhD., Principal Investigator — Department of Surgery, Breast Cancer Center,Inje University Paik Hospital, South Korea
Locations (1):
- Department of Surgery, Breast Cancer Center, Inje University Paik Hospital, Seoul, South Korea